CLINICAL TRIAL: NCT01295229
Title: Feasibility, Efficacy, and Mechanisms of Surgical vs Medical Diabetes Treatment
Brief Title: Calorie Reduction Or Surgery: Seeking Remission for Obesity And Diabetes
Acronym: CROSSROADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kaiser Permanente (Other); Fred Hutchinson Cancer Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David Flum, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 194279; 1R01DK089528-01 (NIH)
Record Dates: First submitted 2011-02-02; First posted 2011-02-14 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Bariatric Surgery; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Intervention (Active Comparator)
  Interventions: Behavioral: Lifestyle Intervention
- Surgery (Active Comparator)
  Interventions: Procedure: laparoscopic Roux-en-Y gastric bypass (RYGB) procedure

INTERVENTIONS:
Procedure: laparoscopic Roux-en-Y gastric bypass (RYGB) procedure — The laparoscopic Roux-en-Y gastric bypass (RYGB) procedure is the most commonly performed bariatric procedure in the United States. Patients randomized to the surgical arm will undergo a standard laparoscopic proximal RYGB, as commonly practiced by GH surgeons, using a 90-cm alimentary limb, 50-cm biliopancreatic limb, antecolic/antegastric approach, and totally stapled technique.
  Other Names: weight loss surgery; bariatric surgery
  Arms: Surgery
Behavioral: Lifestyle Intervention — The lifestyle intervention includes behavior-modification skills counseling combined with training in diet and exercise change. The focus of the exercise intervention is a gradual increase in brisk walking or other activities of similar moderate aerobic intensity. The exercise prescription will consist of at least 45 minutes of exercise, 5 days per week for 12 months. The diet intervention will be conducted by a research dietician with training in behavior modification, with supervision by Dr. Foster-Schubert. In week 1 the dietician will meet for a 60-minute individual session with participants at the FHCRC Prevention Center. Over the next 23 weeks the dietician will conduct one 30-minute group session per week.
  Other Names: Diet and Exercise Program
  Arms: Lifestyle Intervention

SUMMARY:
The escalating pandemics of obesity and type 2 diabetes mellitus (T2DM) are among the most significant contributors to morbidity and mortality worldwide. Roux-en-Y gastric bypass (RYGB) surgery causes profound weight loss and dramatically ameliorates T2DM through mechanisms beyond just weight loss, but its role in diabetes management and the nature of its weight-independent anti-diabetes effects are not well established because of a paucity of appropriate randomized trials, the execution of which is hindered by numerous obstacles. The investigators therefore propose a feasibility study to demonstrate our capacity to identify, recruit, randomize, and track outcomes for 40 adult Group Health members identified as having T2DM and a BMI between 30-40 kg/m2.

DETAILED DESCRIPTION:
The overall goal of the research study is to demonstrate our capacity to identify, recruit, randomize, and track outcomes for 40 adult Group Health members identified as having T2DM and a BMI between 30-40 kg/m2.

Our cohort recruitment strategy will utilize the GH administrative and clinical databases to identify patients with T2DM and a BMI of 30-40 kg/m2. Sufficient numbers (N=4,000) of these individuals will be mailed and surveyed to identify the small minority without strong preferences regarding medical vs. surgical diabetes/obesity treatment. This subset will be invited to become better informed about both strategies using a novel, standardized patient decision aid for shared decision making (SDM) related to bariatric surgery: a high-quality educational video that provides balanced and frequently updated information about the risks and benefits of surgical and non-surgical care. After viewing SDM tool, potential subjects' "willingness to randomize" will be assessed, and a subset of willing patients will actually undergo randomization to either RYGB or a state-of-the-art intensive but reproducible medical/lifestyle intervention.

Forty patients will be randomized to either RYGB or an intensive medical/lifestyle intervention. Twenty members will be randomly assigned to intensive behavioral/medical treatment, and twenty will be randomly assigned to receive gastric bypass surgery. In the non-surgical group, the investigators will study the feasibility and resources needed to deploy a state-of-the-art intensive behavioral intervention to promote weight loss, which includes dietary and exercise components. It will be coupled with diabetes pharmacotherapy treatment consistent with Group Health Clinical Practice Guidelines (http://incontext.ghc.org/clinical/clin_topics/diabetes2/dm2_poc.html).

Patients randomized to the surgical arm will undergo a standard laparoscopic proximal RYGB, as commonly practiced by GH surgeons. The operation and post-operative care will be performed at GH by Dr. Steven Bock, Dr. Jeffery Lander, and their clinical staff, including a team of nutritionists and a Registered Nurse Case Manager who coordinates the care of patients in the GH Bariatric Surgery Program. Surgical patients will also undergo a standardized 8-week pre-operative and 10-month post-operative behavioral treatment regimen with the GH Bariatric Surgery Program.

Participants will have follow-up research visits at 3, 6, 9, and 12 months after randomization, where they will have the following measurements: standardized physically exam by Dr. Foster-Schubert; weight, waist and hip circumferences; systolic and diastolic blood pressure; resting 1-minute pulse; and fasting (12-hour) blood (50 ml) collection.

ELIGIBILITY:
Inclusion Criteria:

* currently enrolled at Group Health
* currently enrolled in a GH insurance product that provides coverage for laparoscopic gastric bypass (e.g., Medicare, PEBB, or has GH bariatric coverage rider)
* age on January 1, 2011 will be between 25 and 65 years
* Diabetes: must meet one or more of the following criteria during the past two years (10/1/08 - 9/30/10):

  1. 1+ fills for a diabetes-specific medication (oral or insulin)
  2. Hemoglobin A1c ≥7.0% on one or more occasions
  3. Fasting Blood glucose ≥126 mg/dL on two or more occasions [separate days]
  4. Random glucose ≥200 mg/dl on two or more occasions [separate days]
  5. One fasting blood glucose ≥126 mg/dL plus one random glucose ≥200 mg/dl [must occur on separate days]
  6. One or more inpatient (primary or secondary hospital discharge) code related to diabetes. See list below.
  7. Two or more outpatient ICD-9 codes related to diabetes (ambulatory visits (AV) only - not telephone, email, emergency department, lab, radiology, or other (IS, OE) encounter types) [Two visits must occur on separate days]
* Obesity: All patients must have a body mass index [BMI] between 30 and <40kg/m2; weight measurement must be within the past two years (10/1/08 - 9/30/10)

Exclusion Criteria:

* Pregnancy within the past one year (10/1/09 - 9/30/10)
* Excluded if the following conditions are recorded within the past two years (10/1/08 - 9/30/10):

  1. malignant tumor
  2. ascites
  3. peritoneal effusion
  4. cirrhosis
  5. schizophrenia
  6. schizoaffective disorder
  7. bipolar disorder
  8. dementia
  9. HIV
  10. inflammatory bowel disease
  11. dialysis
* Exclude if occurred between 1/1/95 - 9/30/10:

  1. Any prior bariatric or major gastrointestinal operation
  2. Any prior liver, heart, intestinal, and/or lung transplant

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Feasibility | April 2011 - January 2012
  Explore the feasibility of a set of novel methods to create an appropriate randomization cohort of patients with type 2 diabetes mellitus (T2DM) and a body mass index (BMI) of 30-40 kg/m2 who are willing to be randomized into either roux-en-Y gastric bypass (RYGB) surgery or an intensive medical/lifestyle intervention. This will be assessed by comparing the number of people recruited to the number randomized and subsequently enrolled in the study.

SECONDARY OUTCOMES:
Efficacy and Mechanisms | April 2011-April 2013
  Participants will complete research visits at Baseline, 6-month and 12-month. Both intervention groups (surgery and lifestyle) will complete the same physical assessments to compare success of the intervention. Physical measures include a fasting blood draw, DEXA scan, exercise treadmill test, anthropometric measures and vitals. Additionally, a subset of participants will be assessed for changes in their immune system before and after the intervention. Measures include an adiopose tissue biopsy and an Oral Glucose Tolerance Test.

CONTACTS AND LOCATIONS:
Overall Officials: David E Cummings, MD, Principal Investigator — University of Washington; David R Flum, MD, MPH, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Group Health Research Institute, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Banerjee S, Garrison LP Jr, Flum DR, Arterburn DE. Cost and Health Care Utilization Implications of Bariatric Surgery Versus Intensive Lifestyle and Medical Intervention for Type 2 Diabetes. Obesity (Silver Spring). 2017 Sep;25(9):1499-1508. doi: 10.1002/oby.21927. Epub 2017 Jul 19. PMID 28722299
- [Derived] Cummings DE, Arterburn DE, Westbrook EO, Kuzma JN, Stewart SD, Chan CP, Bock SN, Landers JT, Kratz M, Foster-Schubert KE, Flum DR. Gastric bypass surgery vs intensive lifestyle and medical intervention for type 2 diabetes: the CROSSROADS randomised controlled trial. Diabetologia. 2016 May;59(5):945-53. doi: 10.1007/s00125-016-3903-x. Epub 2016 Mar 17. PMID 26983924